CLINICAL TRIAL: NCT02459587
Title: Facilitating Use of the Veterans Crisis Line in High-Risk Patients
Brief Title: Crisis Line Facilitation
Acronym: CLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 14-103
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Suicide; Suicide, Attempted; Hospitals, Psychiatric
Keywords: Self-Injurious Behavior; suicide prevention
MeSH Terms: conditions — Suicide; Suicide, Attempted; Self-Injurious Behavior; Suicide Prevention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crisis Line Facilitation (CLF) (Experimental): Crisis Line Facilitation
  Interventions: Behavioral: Crisis Line Facilitation (CLF)
- Enhanced Usual Care (EUC) (Placebo Comparator): Enhanced Usual Care
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Crisis Line Facilitation (CLF) — This single session therapist-delivered intervention addresses Veterans' perceived barriers and facilitators of crisis line use during periods of suicidal crisis. The CLF session culminates with the Veteran calling the Crisis Line with the therapist in the room as a way for the Veteran to practice the logistics of making the call and to have direct experiences that may counter any negative beliefs about Crisis Line use.
  Arms: Crisis Line Facilitation (CLF)
Behavioral: Enhanced Usual Care (EUC) — Those in the EUC condition received the same promotional items and information about the Veterans Crisis Line (VCL) as the CLF condition. Participants were encouraged to seek help via a provider or the VCL if they felt suicidal in the future. Research staff briefly explained key information about the VCL to those in the EUC condition (e.g., the links between the VCL and the VA, the 24/7/365 availability, etc.).
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
This study is a randomized controlled trial (n = 301) of a new single-session intervention, called Crisis Line Facilitation (CLF), compared to an enhanced usual care condition on utilization of the Veterans Crisis Line and other mental health services as well as suicide attempt(s). All participants were recruited during an inpatient psychiatric stay for the treatment of a recent suicidal crisis and will be re-assessed at 3-, 6- and 12-months post baseline. If successful, the proposed study will provide key data on the potential efficacy of a brief tool to improve the utilization of an existing resource, the Veterans Crisis Line, to reduce suicidal behaviors in VHA patients.

DETAILED DESCRIPTION:
Veterans Health Administration (VHA) patients are at a significantly elevated risk for fatal and non-fatal suicide attempts and identifying strategies to reduce the risk of suicidal behavior among members of the military and Veterans is a high national priority. The VHA has invested extensively in suicide prevention and, as part of these efforts; the Veterans Crisis Line was developed as an important resource for Veterans and their families. Utilization of the Veterans Crisis Line has expanded steadily since it first opened and, currently, it receives over 20,000 calls per month. Despite high utilization of the Crisis Line, no data are currently available on whether use of the Veterans Crisis Line reduces an individual's likelihood of a suicide attempt or death and it is not feasible to test the efficacy of the Crisis Line in a randomized controlled trial because it is nationally available to all Veterans and their families. More importantly, the Veterans Crisis Line may not reach those individuals at most acute risk for suicide. The investigators' study team conducted a small survey of Veterans treated for recent suicidal crisis in a VHA inpatient psychiatric unit and found that less than half had ever utilized the Veterans Crisis Line and less than a third had used it within the past year. Consequently, the investigators have developed and gathered pilot data on a brief intervention designed to increase utilization of the Veterans Crisis Line among high risk patients, called Crisis Line Facilitation (CLF). This single-session intervention involves a discussion of the patient's perceived barriers of crisis line use during periods of suicidal crisis. The CLF session ends with the patient calling the Crisis Line with the therapist in the room as a way for Veterans to practice the logistics of making the call and to have direct experiences that may counter any negative beliefs about Veterans Crisis Line use. This study recruited 301 participants who were treated for a suicidal crisis in VHA inpatient psychiatric but had not recently used the Veterans Crisis Line. This study is a randomized controlled trial of the impact of CLF compared to enhanced usual care (EUC) on utilization of the Veterans Crisis Line and other mental health services as well as suicide attempt(s). All participants will be re-assessed at 3-, 6- and 12-months post baseline. Analyses will also examine the extent to which post-baseline Crisis Line use mediates the effect of random assignment to CLF on subsequent suicidal behaviors. Qualitative interviews at the end of the study will help understand barriers and facilitators of future implementation of the CLF intervention. If successful, the proposed study will provide key data on the potential efficacy of a brief intervention to improve the utilization of an existing resource, the Veterans Crisis Line, to reduce suicidal behaviors in VHA patients. Developing a brief and effective approach to encourage use of the Crisis Line has the potential to have a significant and substantial impact on suicide rates within the VHA and could be modified and exported to other populations and settings.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for screening (Part 1).

* adults age 18 years of age or older receiving care in an inpatient psychiatric unit at either the BC VAMC or AA VAMC;
* mention of a significant suicidal crisis within the intake note;
* medically stable and able to provide informed consent; and
* Mini-Mental State Examination (MMSE) score greater than or equal to 21.

Additional inclusion criteria for the full randomized study (Part 2):

* no reported use of the Veterans Crisis Line within the past 12-months;
* report current suicidal ideation (BSS greater than or equals 5 during the week prior to hospitalization) as reported during the screening interview.

Exclusion Criteria:

Exclusion criteria for screening and full study:

* patients who do not understand English;
* prisoners;
* patients deemed unable to provide informed consent as stated above;
* patients who recently received or are scheduled to receive electroconvulsive therapy (ECT); and
* profound psychotic symptoms and/or cognitive deficits that would prevent patients from understanding the content of the intervention and/or assessments.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Ilgen, PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Battle Creek VA Medical Center, Battle Creek, MI, Battle Creek, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Crisis Line Facilitation: Crisis Line Facilitation (CLF) is a single-session intervention which focuses on increasing awareness and motivation to contact the Veterans Crisis Line during a suicidal crisis.
- Enhanced Usual Care: Enhanced Usual Care (EUC) provided educational materials about the Veterans Crisis Line in addition to the standard of care provided on the inpatient hospital unit.
Period: 3-Month Follow-up Assessment
Arm/Group | Crisis Line Facilitation | Enhanced Usual Care
Started | 157 | 150
Completed | 125 | 119
Not Completed | 32 | 31
Not completed — Death | 0 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 27 | 22
Not completed — Researcher withdrew | 2 | 4
Period: 6-month Follow-up Assessment
Arm/Group | Crisis Line Facilitation | Enhanced Usual Care
Started | 152 (Total excludes participants who withdrew participation or were deceased prior to follow-up.) | 141 (Total excludes participants who withdrew participation or were deceased prior to follow-up.)
Completed | 128 | 116
Not Completed | 24 | 25
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 21 | 22
Period: 12-month Follow-up Assessment
Arm/Group | Crisis Line Facilitation | Enhanced Usual Care
Started | 149 (Total excludes participants who withdrew participation or were deceased prior to follow-up.) | 138 (Total excludes participants who withdrew participation or were deceased prior to follow-up.)
Completed | 127 | 111
Not Completed | 22 | 27
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 18 | 22
Not completed — Researcher withdrew | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crisis Line Facilitation | Enhanced Usual Care | Total
Number analyzed (Participants) | 157 | 150 | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.2 (12.8) | 46.8 (13.5) | 47.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 138 | 130 | 268
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 22 | 54
  White | 112 | 113 | 225
  More than one race | 7 | 9 | 16
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 157 | 150 | 307
Columbia Suicide Severity Scale (C-SSRS): Most severe suicidal ideation, Lifetime [Count of Participants; unit: Participants]
  No suicidal ideation | 5 | 1 | 6
  Wish to be dead / Non-Specific Active Suicidal Thoughts | 20 | 15 | 35
  Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act | 17 | 24 | 41
  Active Suicidal Ideation with Some Intent to Act, without Specific Plan | 23 | 21 | 44
  Active Suicidal Ideation with Specific Plan and Intent | 92 | 89 | 181
Columbia Suicide Severity Scale (C-SSRS): Lifetime Suicide Attempts [Count of Participants; unit: Participants]
  No attempts | 46 | 41 | 87
  One attempt | 31 | 37 | 68
  2 or more attempts | 80 | 72 | 152
Utilization of the Veterans Crisis Line, Lifetime [Count of Participants; unit: Participants] — For participants who endorsed contacting the VCL in their lifetime, these contacts were not within the previous 12 months.
  Participants
    Never contacted VCL | 104 | 104 | 208
    Contacted VCL once | 25 | 22 | 47
    Contacted VCL 2 or more times | 28 | 24 | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Veterans Crisis Line (VCL) Contact Events Per Days at Risk
Description: The primary data source for information regarding use of the VCL was collected via researcher-administered interview questions during the TimeLine Follow Back assessment. Participants were asked to recall how many times since the last assessment in which they contacted the VCL for any reason. For contacts that occurred, participants were asked to recall the date of these contacts and the type of contact that was made (e.g. phone call, text, or chat).
Time Frame: 1 year
Population: Analytical sample consists of participants who completed at least one follow-up.
Measure: Number; unit: VCL Contact Events
Units Other Than Participants: Person-days
Arm/Group | Crisis Line Facilitation | Enhanced Usual Care
Number analyzed (Participants) | 141 | 131
Number analyzed (Person-days) | 50488 | 44194
VCL Contact Events | 48 | 35
Statistical Analysis 1: Comparison: Crisis Line Facilitation vs Enhanced Usual Care; Test type: Superiority — Survival analysis using start/stop counting method to identify time until event, structured to allow for multiple events per person. VCL contacts with and without suicide ideation were combined, due to low counts; p = 0.33, Regression, Cox — 2-tailed P-value above was calculated from type III test; Model was structured to allow multiple events per person. No covariates; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.80 to 1.92], Standard Error of Mean 0.222 — Model was structured to allow multiple events per person. No covariates. HR based on parameter estimate = -0.218 (SEM=0.222)

2. Secondary Outcome: Number of Suicide Behavior Events Per Days at Risk
Description: The primary data source for suicidal behaviors was the TimeLine Follow Back, a semi-structured researcher-administered interview. Participants were asked to report actual, interrupted, and aborted attempt events that occurred since the last study assessment. Definitions for these events were derived from the Columbia Suicide Severity Rating Scale (C-SSRS) Suicidal Behaviors subsection [also administered during the assessment], and dates for these events were entered into the TimeLine Follow Back.
Time Frame: 1 year
Population: Analytical sample consists of participants who completed at least one follow-up.
Measure: Number; unit: Suicide Behavior Events
Units Other Than Participants: Person-days
Arm/Group | Crisis Line Facilitation | Enhanced Usual Care
Number analyzed (Participants) | 141 | 131
Number analyzed (Person-days) | 50485 | 44192
Suicide Behavior Events | 67 | 116
Statistical Analysis 1: Comparison: Crisis Line Facilitation vs Enhanced Usual Care; Test type: Superiority — Survival analysis using start/stop counting method to identify time until event, structured to allow for multiple events per person; p < 0.0001, Regression, Cox — All tests of significance were 2-tailed. P-value above is type III. No covariates; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.38 to 0.70], Standard Error of Mean 0.153 — Cox Proportional Hazards Model was structured to allow multiple events per person. No covariates. HR based on parameter estimate = -0.660 (SEM=0.153)

3. Secondary Outcome: Outpatient General Mental Health Clinic Visit
Description: The primary data source for general mental health treatment service utilization was a modified version of the Treatment Services Review, an researcher-administered structured interview. Participants were asked to report whether or not they had been to a mental health clinic for therapy or medications since the last study assessment.
Time Frame: 1 year
Population: Analytical sample consists of participants who completed at least one follow-up.
Measure: Mean (Standard Deviation); unit: Mean number of visits
Arm/Group | Crisis Line Facilitation | Enhanced Usual Care
Number analyzed (Participants) | 141 | 131
Mean number of visits | 24.5 (25.2) | 21.2 (20.7)
Statistical Analysis 1: Comparison: Crisis Line Facilitation vs Enhanced Usual Care; Test type: Superiority — Two binary variables were derived from Treatment Services Review responses to identify any general mental health service utilization, one binary variable for Baseline and another for any outpatient mental health service utilization at any time point in the 1 year follow-up period. The Baseline variable was included as a main-effects covariate; p = 0.66, Regression, Logistic; Bivariate logistic, adjusted for (1) if any general outpatient mental heath visits at baseline (0) otherwise; Odds Ratio, log = 1.146, 95% CI 2-sided [0.604 to 2.176]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious adverse events were death and other life-threatening events. Adverse events were suicidal ideation or behaviors, breach of confidentiality, hospitalizations or other interventions resulting from suicidal thoughts, behaviors, or substance use (e.g. overdose, acute intoxication), hospitalizations for medical reasons, accidents or injuries (including non-suicidal self-injury), and discomfort associated with answering difficult questions.
Arm/Group | Crisis Line Facilitation | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 4/157 | 3/150
Serious Adverse Events (participants affected / at risk) | 4/157 | 7/150
Other Adverse Events (participants affected / at risk) | 91/157 | 97/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crisis Line Facilitation (N=157) | Enhanced Usual Care (N=150)
Death by heart attack (Cardiac disorders) | 0 (0) | 1 (1)
Death by suicide (Psychiatric disorders) | 2 (2) | 2 (2)
Death by overdose (Psychiatric disorders) | 2 (2) | 0 (0)
Hospitalization (Psychiatric disorders) | 0 (0) | 4 (4) — Participant inpatient hospitalization for to a suicide or substance related reason immediately following a study interaction
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Crisis Line Facilitation (N=157) | Enhanced Usual Care (N=150)
Psychiatric Hospitalization: Suicidal Ideation (Psychiatric disorders) | 42/155 (74) | 40 (74)
Medical Hospitalization (Surgical and medical procedures) | 8 (11) | 18 (23) — Includes hospitalizations for medical related events only (e.g. surgery, accidents, injuries, illnesses)
Residential Treatment (Psychiatric disorders) | 44 (53) | 33 (38) — Treatment for psychiatric or substance use disorders
Suicide Attempt (Psychiatric disorders) | 19 (36) | 20 (26)
Psychiatric Hospitalization: Acute Substance Use (Psychiatric disorders) | 9 (10) | 6 (9) — Includes hospitalizations for detoxification, intoxication, overdose, or increased substance use.
Psychiatric Hospitalization: General (Psychiatric disorders) | 6 (8) | 12 (15) — Includes hospitalizations for general mental health reasons, excluding suicidal ideation or substance use

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Ann Arbor (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT02459587/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Battle Creek (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT02459587/Prot_SAP_001.pdf
  • Informed Consent Form: Main Study Consent (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT02459587/ICF_002.pdf
  • Informed Consent Form: Qualitative Interview Consents (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT02459587/ICF_003.pdf